CLINICAL TRIAL: NCT03500354
Title: Nutritional Drink in Gastroparesis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to another institution and closed the study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00157677
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2022-03

CONDITIONS: Gastroparesis
Keywords: malnutrition
MeSH Terms: conditions — Gastroparesis; Malnutrition

STUDY DESIGN:
Intervention Model Description: Pilot feasibility open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrient (Experimental): Nutrient drink
  Interventions: Dietary Supplement: Nutrient drink

INTERVENTIONS:
Dietary Supplement: Nutrient drink — High calorie drink with therapeutic supplements

SUMMARY:
Gastroparesis is a chronic, morbid and costly neuromuscular disorder of the stomach characterized by delayed gastric emptying in the absence of gross structural abnormalities. The periprandial symptoms associated with this disease can preclude adequate oral intake and often lead to weight loss and nutritional deficiencies 1. These manifestations are largely due to impaired gastric accommodation of meals and delayed transfer of food boluses from the stomach into the duodenum2. Consequently, the investigators hypothesize that dietary supplementation with a low volume, hypercaloric nutritional drink can help prevent malnutrition, decrease symptom burden and improve health-related quality of life in this population. Due to the paucity of such a supplement, the investigators developed a novel nutritional drink designed to maximize tolerability in patients with gastroparesis . This nutritional drink was tested on healthy volunteers (phase I) and passed the palatability test. The investigators now aim to test the tolerability of this drink on gastroparesis patients.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the safety and tolerability of the nutritional drink in gastroparesis patients.

Secondary objective:

To evaluate the efficacy of the nutritional drink in gastroparesis patients.

Study Procedures This study will be a pilot, open-label, trial in gastroparesis patients. A total of 20 patients will be recruited from the gastroenterology gastroparesis clinic. If the volunteer meets eligibility criteria, a co-investigator will contact the patient to schedule a study visit with a nutritionist and obtain a written consent. The contact and screening information of patients that are successfully recruited will be documented, placed in the participant's study folder and stored in a locked cabinet in the research unit. Any information documented during the screening process for patients who do not meet basic eligibility criteria or do not wish to participate will be immediately destroyed.

Patients will be given enough supply of the nutrition drink for (4 weeks) and asked to consume 200 ml of the drink three times daily. A follow-up call will be scheduled on day 2, day 7 and at the end of the study to make sure patients are tolerating the drink. Participants will be allowed to consume water and food as desired during the study period but will need to maintain an accurate food diary for at least one week prior to enrollment and during the study (at 2 weeks and at 4 weeks) along with weight measurements at baseline, 2 weeks, 4 weeks and 6 weeks. The participants will be asked to complete a palatability questionnaire. They will also complete the Gastroparesis Cardinal Symptom Index (GCSI) daily diary and the PROMISE scale prior to enrollment as a baseline for their symptoms and again at 2 weeks, 4 weeks (end of the study) and 6 weeks. Changes in these scales from baseline will determine the efficacy and possibly side effects of the nutritional drink.

Study duration and number of study visits required of research participants:

4 weeks, initial study visit with a nutritionist for screening and consenting followed by 3 follow-up phone calls on day 2, day 7 and at 4 weeks (the end of the study) and a final study visit at 6 weeks (2 weeks after finishing the study)

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastroparesis confirmed with symptoms and a gastric emptying study.
* Inability to maintain adequate caloric intake by standard dietary measures for gastroparesis due to gastrointestinal symptoms

Exclusion Criteria:

* Recent diagnosis of disorder other than gastroparesis that could affect food intake
* Oropharyngeal dysphagia or other condition with risk for aspiration from oral ingestion.
* Allergic reactions to any of the ingredients of the nutritional drink
* Current pregnancy. Pregnancy status will be determined by questioning the potential subject.
* Patient with gastrostomy/jejunostomy tube feeds or on total parenteral nutrition
* Currently taking any anti-coagulant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female or male
Enrollment: 0 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Tolerability will be measured by the Palatability Questionnaire at 2 days | 2 days post-intervention
  Patients will be given enough supply of the nutrition drink for 4 weeks and asked to consume 200 ml of the drink three times daily. A follow-up call will be scheduled on day 2 of the study to make sure patients are tolerating the drink.
  Tolerability will be measured by the Palatability Questionnaire which rates six items on a scale of 1 to 5 (1= strongly disagree and 5= strongly agree. The six items are:
  * The formula/supplement tasted very good.
  * The formula/supplement tasted very bad.
  * I had no problems drinking the supplement.
  * Drinking the supplement made me feel ill.
  * I could drink more of this supplement anytime
  * I would never drink more of this supplement again
Tolerability will be measured by the Palatability Questionnaire at 7 days | 7 days post-intervention
  Patients will be given enough supply of the nutrition drink for 4 weeks and asked to consume 200 ml of the drink three times daily. A follow-up call will be scheduled on day 7 of the study to make sure patients are tolerating the drink.
  Tolerability will be measured by the Palatability Questionnaire which rates six items on a scale of 1 to 5 (1= strongly disagree and 5= strongly agree. The six items are:
  * The formula/supplement tasted very good.
  * The formula/supplement tasted very bad.
  * I had no problems drinking the supplement.
  * Drinking the supplement made me feel ill.
  * I could drink more of this supplement anytime
  * I would never drink more of this supplement again
Tolerability will be measured by the Palatability Questionnaire at 4 weeks | 4 weeks post-intervention
  Patients will be given enough supply of the nutrition drink for 4 weeks and asked to consume 200 ml of the drink three times daily. A follow-up call will be scheduled at 4 weeks to make sure patients are tolerating the drink.
  Tolerability will be measured by the Palatability Questionnaire which rates six items on a scale of 1 to 5 (1= strongly disagree and 5= strongly agree. The six items are:
  * The formula/supplement tasted very good.
  * The formula/supplement tasted very bad.
  * I had no problems drinking the supplement.
  * Drinking the supplement made me feel ill.
  * I could drink more of this supplement anytime
  * I would never drink more of this supplement again
Safety will be measured by the NIH PROMISE scale at baseline | Baseline
  This will be measured by the NIH PROMISE scale. This is a 10 point scale (0=none and 10= most severe) that rates the following symptoms:
  * Pain, especially in the abdomen, chest or back
  * Abdominal distension (bloating, sensation of excess gas)
  * Difficulty eating, sensation of food being stuck in the stomach.
  * Difficulty with bowel movements (constipation or straining)
  * Nausea and/or vomiting
  * Thirst
  * Weakness, lack of energy, fatigue, difficulty moving.
Safety will be measured by the NIH PROMISE scale at 2 weeks | 2 weeks post-intervention
  This will be measured by the NIH PROMISE scale. This is a 10 point scale (0=none and 10= most severe) that rates the following symptoms:
  * Pain, especially in the abdomen, chest or back
  * Abdominal distension (bloating, sensation of excess gas)
  * Difficulty eating, sensation of food being stuck in the stomach.
  * Difficulty with bowel movements (constipation or straining)
  * Nausea and/or vomiting
  * Thirst
  * Weakness, lack of energy, fatigue, difficulty moving.
Safety will be measured by the NIH PROMISE scale at 4 weeks | 4 weeks post-intervention
  This will be measured by the NIH PROMISE scale. This is a 10 point scale (0=none and 10= most severe) that rates the following symptoms:
  * Pain, especially in the abdomen, chest or back
  * Abdominal distension (bloating, sensation of excess gas)
  * Difficulty eating, sensation of food being stuck in the stomach.
  * Difficulty with bowel movements (constipation or straining)
  * Nausea and/or vomiting
  * Thirst
  * Weakness, lack of energy, fatigue, difficulty moving.
Safety will be measured by the NIH PROMISE scale at 6 weeks | 6 weeks post-intervention
  This will be measured by the NIH PROMISE scale. This is a 10 point scale (0=none and 10= most severe) that rates the following symptoms:
  * Pain, especially in the abdomen, chest or back
  * Abdominal distension (bloating, sensation of excess gas)
  * Difficulty eating, sensation of food being stuck in the stomach.
  * Difficulty with bowel movements (constipation or straining)
  * Nausea and/or vomiting
  * Thirst
  * Weakness, lack of energy, fatigue, difficulty moving.

SECONDARY OUTCOMES:
Improvement in gastroparesis symptoms | Baseline, 2, 4 and 6 weeks
  Change in weight compared to baseline
Improvement in gastroparesis symptoms | Baseline, 2, 4 and 6 weeks
  Changes in the Gastroparesis Cardinal Symptom Index (GCSI) daily diary as compared to baseline. This is a six point severity scale (0-5 with 0= none and 5 = very severe) that rates the following symptoms
  * Nausea
  * Early satiety
  * Postprandial fullness
  * Bloating
  * Upper abdominal pain
  * Retching
  * Vomiting
  * Stomach fullness
  * Loss of appetite
  * Stomach or belly visibly large

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj J Pasricha, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No